CLINICAL TRIAL: NCT02767037
Title: SudoScan as a Biomarker of Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Ron Postuma, Neurologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MP-CUSM-15-472
Record Dates: First submitted 2016-01-22; First posted 2016-05-10 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Parkinson's disease (PD) patients (Active Comparator): 40 patients will be recruited. All will meet criteria for probable PD, according to the new MDS Clinical Diagnostic criteria. All participants will be 40 or older (young-onset PD includes many genetic causes, which often have normal autonomic function).
  Interventions: Device: Sudoscan and clinical assessment; Genetic: Skin biopsy
- parkinsonsism (non-PD) patients (Active Comparator): 20 patients will also be recruited. These will include patients with progressive supranuclear palsy, multiple system atrophy, 'vascular parkinsonism' or corticobasal syndrome. All patients will have parkinsonism according to UK brain bank criteria, with a diagnosis of one of the above conditions made according to gold-standard expert evaluation. No patient will meet MDS Criteria for probable PD.
  Interventions: Device: Sudoscan and clinical assessment; Genetic: Skin biopsy
- idiopathic REM sleep behavior disorder patient (Active Comparator): 40 patients will be recruited. All patients will have polysomnogram-confirmed RBD according to American Academy of Sleep Medicine Criteria. Patients will be free of parkinsonism and dementia according to neurological examination and will have no untreated sleep apnea, epilepsy, or other abnormalities that could cause dream enactment behavior.
  Interventions: Device: Sudoscan and clinical assessment; Genetic: Skin biopsy
- Controls (Placebo Comparator): 40 controls will be age matched (within 5 years) and sex-matched (with >90% concordance). All controls will have an examination confirming the absence of parkinsonism, and will have no symptoms of REM sleep behavior disorder, as assessed with the RBD1Q and expert interview.
  Interventions: Device: Sudoscan and clinical assessment; Genetic: Skin biopsy

INTERVENTIONS:
Device: Sudoscan and clinical assessment — The primary variable will be electrochemical skin conductance (ESC), as assessed by the SudoScan (Impeto Medical, France). The clinical assessment will include a neurological evaluation (including MDS-UPDRS), evaluation of autonomic symptoms and signs, EKG, evaluation of possible neuropathy and evaluation of non-motor variables.
Genetic: Skin biopsy — Evaluation of the denervation and synuclein deposition of skin biopsy

SUMMARY:
Currently, there is no clear diagnostic test that can be used to confirm the diagnosis of Parkinson's disease, or a biomarker that can track its progression. Patients with Parkinson's have many abnormalities of the autonomic nervous system, which may be related to Parkinson's changes outside of the brain. A new device called the SudoScan, which measures autonomic sweating changes, may be a simple way to test for autonomic changes in Parkinson's.

The investigator plan to see whether SudoScan can identify Parkinson's disease and whether SudoScan abnormalities might be present even in early (prodromal) Parkinson's stages.

The investigator will assess SudoScan in a group of Parkinson's patients, normal healthy controls, patients with non-Parkinson's neurodegeneration, and patients with REM sleep behavior disorder (an early/prodromal Parkinson's state). Abnormalities will be correlated with standard autonomic tests and with skin biopsy findings Parkinson's degeneration in the peripheral autonomic fibers.

If the investigator can find a reliable way to diagnose and follow Parkinson's disease, he will be able to correctly identify Parkinson's (even in its earliest stages). This will improve the chance to find protective treatments against Parkinson's, by preventing false diagnosis and by providing a new marker to track disease progression.

If successful, the investigator will aim to validate the findings on a large sample of Parkinson's and also to track changes over time in the original cohorts

ELIGIBILITY:
Inclusion Criteria:

1. PD patients: All will meet criteria for probable PD, according to the new MDS Clinical Diagnostic criteria
2. Non-PD parkinsonism patients: They will have with progressive supranuclear palsy, multiple system atrophy, 'vascular parkinsonism' or corticobasal syndrome. All patients will have parkinsonism according to UK brain bank criteria, with a diagnosis of one of the above conditions made according to gold-standard expert evaluation. No patient will meet MDS Criteria for probable PD.
3. iRBD patients: All patients will have polysomnogram-confirmed RBD according to American Academy of Sleep Medicine Criteria. Patients will be free of parkinsonism and dementia according to neurological examination and will have no untreated sleep apnea, epilepsy, or other abnormalities that could cause dream enactment behavior.
4. Controls: These will be age matched (within 5 years) and sex-matched (with >90% concordance). All controls will have an examination confirming the absence of parkinsonism, and will have no symptoms of REM sleep behavior disorder, as assessed with the RBD1Q and expert interview.

Exclusion Criteria:

1. Diabetes Mellitus - In addition to causing autonomic neuropathy, hyperglycemia itself is known to interfere with results of the sudomotor scan
2. Any preceding diagnosis of autonomic neuropathy (of a cause other than PD)
3. Dementia of severity sufficient to preclude informed consent, MoCA <23.
4. Prescription of medications that directly alter peripheral autonomic function, including beta-blockers, sympatholytics (i.e. clonidine) and non-specific alpha-blockers.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Electrochemical skin conductance | up to 6 months

SECONDARY OUTCOMES:
PD severity-Hoehn and Yahr stage | up to 6 months
  PD severity will be assessed with the Hoehn and Yahr
PD severity-MDS-UPDRS | up to 6 months
  PD severity will be assessed with the MDS-UPDRS
Autonomic symptoms and signs | up to 6 months
EKG | up to 6 months
  Cardiac autonomic denervation will be assessed with analysis of heart rate variability on EKG
Neuropathy | up to 6 months
  Patients will be screened for neuropathy with the 5-item peripheral neuropathy screening interview
Non-motor symptoms associated with PD | up to 6 months
  Non-motor variables with be assessed with Parts I and II of the MDS-UPDRS
Skin biopsy | up to 12 months
  Denervation and synuclein deposition of skin biopsy will include staining for proteinase-k-resistant synuclein (5C12 antibody) and neuronal markers to determine density of peripheral innervation

IPD SHARING:
Plan to Share IPD: Yes
De-identified clinical data will be shared with the Michael J. Fox Foundation (the study funder) for Parkinson's research. These data may be kept for storage at a central repository either hosted by the Michael J. Fox Foundation, its collaborators, or consultants and will be kept indefinitely. In order to advance scientific discoveries, your de-identified data will be made publically available (with no personal identifying information) for the intended use of research in Parkinson's disease as well as other biomedical research studies that may not be related to Parkinson's disease.